CLINICAL TRIAL: NCT04000945
Title: Evaluation of Safety and Efficacy of the BTL-899 Device for Non-invasive Lipolysis and Circumference Reduction of Abdomen When Compared to a Sham Treatment
Brief Title: Effect of the BTL-899 Therapy for Non-invasive Lipolysis and Circumference Reduction of Abdomen When Compared to a Sham Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BTL-899S
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Improvement of Abdomen Appearance

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BTL-899 Therapy Arm (Experimental)
  Interventions: Device: BTL-899
- Sham Arm (Sham Comparator)
  Interventions: Device: Sham

INTERVENTIONS:
Device: BTL-899 — Treatment with BTL-899 device, 3 therapies
  Arms: BTL-899 Therapy Arm
Device: Sham — Sham treatment with BTL-899 device, 3 visits
  Arms: Sham Arm

SUMMARY:
The study is a prospective single-blinded two-arms study that includes three treatment procedures and four follow-up visits

DETAILED DESCRIPTION:
This study will evaluate the clinical efficacy and safety of the BTL-899 device for non-invasive lipolysis and circumference reduction of abdomen. The study is a prospective single-blinded two-arms study. The subjects will be enrolled and assigned into a two study groups. All subjects will complete three (3) treatment visits and will be invited to four (4) follow-up visits 1, 2, 3 and 6-months after the final treatment. 6-months follow-up visit is the optional one.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years
* Voluntarily signed informed consent form
* BMI ≤ 35 kg/m2
* Women of child-bearing potential are required to use birth control measures during the whole duration of the study
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring during study participation
* Subjects willing and able to maintain his/her regular (pre-procedure) diet and exercise regimen without effecting significant change in either direction during study participation

Exclusion Criteria:

* Cardiac pacemakers
* Cardiovascular diseases
* Implanted defibrillators, implanted neurostimulators
* Electronic implants
* Disturbance of temperature or pain perception
* Pulmonary insufficiency
* Metal implants
* Drug pumps
* Malignant tumor
* Hemorrhagic conditions
* Septic conditions and empyema
* Acute inflammations
* Systemic or local infection such as osteomyelitis and tuberculosis
* Contageous skin disease
* Elevated body temperature
* Pregnancy
* Breastfeeding
* Injured or otherwise impaired muscles
* Scars, open lesions and wounds at the treatment area
* Basedow's disease
* Previous liposuction in the treatment area in the last six months
* Abdominal wall diastasis
* Unstable weight within the last 6 months
* Previous body contouring treatments in the abdomen area in the last three months

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-12-03 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the BTL-899 treatment for change in abdominal circumference | 4 months
  Comparison of change in abdominal circumference at the final follow-up visit between two study groups.
Occurrence of adverse events | 7 months
  The occurrence of adverse events will be followed throughout the whole study.

SECONDARY OUTCOMES:
Efficacy of BTL-899 treatment for abdominal fat and circumference reduction, as assessed by two blinded evaluators | 4 months
  Evaluation of aesthetic improvement achieved by abdominal fat and circumference reduction using photographs before and after the treatment.
Efficacy of the BTL-899 treatment for change in abdominal circumference | 4 months
  Comparison of change in abdominal circumference at all study visits after the first therapy between two study groups.
Efficacy of the BTL-899 treatment for abdominal fat reduction | 4 months
  Comparison of fat reduction between two study groups using ultrasound images.
Subject's satisfaction with study treatment | 4 months
  Subject's satisfaction with the therapy results evaluated through the Subject Satisfaction Questionnaire (5-point scale).
Therapy comfort during the study treatment. | 1 month
  Therapy comfort during the treatment evaluated through the Therapy Comfort Questionnaire (10-point scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Dr-Denkova Dermatology, Sofia, Bulgaria